CLINICAL TRIAL: NCT02485405
Title: Gut Permeability in Volunteers Participating in a Stress Test
Brief Title: Gut Permeability and Stress
Acronym: SP15
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Caroline Linninge, PhD, Lund University
Other Study IDs: SP15_CarolineLinninge
Record Dates: First submitted 2015-06-23; First posted 2015-06-30 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Stress
MeSH Terms: interventions — Psychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Saliva Plasma/Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- stressed: stressed volunteers perform Trier social stress test
  Interventions: Other: Trier social stress test
- non-stressed: non-stressed volunteers perform Trier social stress test
  Interventions: Other: Trier social stress test

INTERVENTIONS:
Other: Trier social stress test — Volunteers perform Trier social stress test

SUMMARY:
The purpose of this study is to analyse gut permeability and stress.

DETAILED DESCRIPTION:
Healthy male volunteers (aged 19-35 years) participate in Trier social stress test while saliva and blood samples are withdrawn.

Saliva will be used for analysis of cortisol and blood will be used for analysis of various biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Man, 19-35 years old
* Healthy

Exclusion Criteria:

* Psychological disorders
* Use of antibiotics or other drugs

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy men aged 19-35 years old
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-06; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
gut permeability (marker measured in plasma/serum) in healthy young men participating in Trier social stress test | Volunteers will be followed by one hour after Trier social stress test

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Linninge, PhD, Principal Investigator — Lund University
Locations (1):
- Lund University, Lund, Sweden